CLINICAL TRIAL: NCT06180174
Title: Phase I Clinical Study of CD19-targeting Chimeric Antigen Receptor T Lymphocyte (MC-1-50) Formulation for the Treatment of Relapsed/Refractory CD19-positive B-cell Non-Hodgkin Lymphoma (B-NHL)
Brief Title: Clinical Research of CD19 Targeted CAR-T Cell in Relapsed/Refractory B Cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB10
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: B Cell Lymphoma; Non Hodgkin Lymphoma
Keywords: CAR-T; CD19
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MC-1-50 cell preparation (Experimental): Patients will be be treated with CD19 CAR- T cells
  Interventions: Biological: MC-1-50

INTERVENTIONS:
Biological: MC-1-50 — A single infusion of CD19 CAR-T cells will be administered intravenously after lymphodepletion

SUMMARY:
This is a single-arm, open-label, dose-escalation phase I clinical study to explore the safety, tolerability, and cytokinetic characteristics of MC-1-50 cell formulation, and to preliminarily observe the efficacy of MC-1-50 cell formulation in subjects with relapsed/refractory CD19-positive B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
Based on the specific CD19-targeting CAR-T developed on the PrimeCARTM platform, the cell preparation time is about 3 days, which can greatly shorten the waiting time of patients, improve production efficiency and reduce production costs. At the same time, MC-1-50 products have a high proportion of T naive cells, which can play a therapeutic effect at a very small infusion dose to improve safety. In this study, a "3+3" design was adopted, and four dose groups were set up with 1×105/kg, 3×105/kg, 5×105/kg, and 10×105/kg CAR-positive cells, respectively (the upper limit of the total number of cells was not more than 1×108 CAR-positive cells). All subjects received only one infusion of MC-1-50 cells.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or his/her guardian agrees to participate in the clinical trial and signs the ICF, indicating that he/she understands the purpose and procedure of the clinical trial and is willing to participate in the study;
2. Age ≥18 years old, gender unlimited;
3. Confirmed cytological or histological diagnosis of B-cell non-Hodgkin lymphoma according to WHO 2017 criteria, including the following pathological types:

   1. Diffuse large B-cell lymphoma: including non-specific type (DLBCL, NOS), chronic inflammatory associated DLBCL, primary cutaneous DLBCL (leg type), EBV-positive DLBCL (NOS);
   2. High-grade B-cell lymphomas (including NOS and high-grade B-cell lymphomas with MYC and BCL2 and/or BCL6 rearrangements);
   3. Primary mediastinal large B-cell lymphoma;
   4. Rich T/ histiocytic large B-cell lymphoma;
   5. Transformed DLBCL (e.g., transformed DLBCL of follicular lymphoma, chronic lymphocytic leukemia/small B lymphocytic lymphoma, marginal zone lymphoma, etc.);
   6. Grade 3b follicular lymphoma (FL3b);
4. Have received adequate treatment with CD20 monoclonal antibody and anthracyclines in the past (except for those who are negative for CD20 and anthracyclines, or who are unable to tolerate or adapt to CD20 monoclonal antibody therapy or have other conditions in which the use of CD20 monoclonal antibody is not considered appropriate by the investigators), For those who are allergic to CD20 monoclonal antibody, or have intolerable serious adverse reactions after use, or have active infections and serious cardiovascular problems, etc.), the definition of relapse or refractory is met during screening:

   1. Recurrence: recurrence of disease progression or recurrence after achieving CR with standard treatment;
   2. Difficult to treat: The best curative effect after at least 4 courses of first-line treatment/at least 2 courses of end-line treatment (2 lines and more) is disease stabilization (SD), and the SD maintenance time after the last dose is not more than 6 months; Or the best response to the last treatment was disease progression (PD);
   3. No remission, disease progression or recurrence after autologous hematopoietic stem cell transplantation;
   4. Patients with transformational lymphoma who received chemotherapy prior to transformation and did not go into remission, disease progression, or relapse after salvage therapy after transformation.
5. Immunohistochemical or flow cytometry results showed positive CD19 expression;
6. ECOG 0 ~ 1 points;
7. The expected survival time is 12 weeks or more;
8. According to the 2014 edition of Lugano standard, there is at least one two-dimensional measurable lesion as the evaluation basis: for intranodular lesion, it is defined as: long diameter >1.5cm; For extranodal lesions, the length diameter should be >1.0cm;
9. The functions of important organs are basically normal:

   1. Cardiac function: cardiac echocardiography suggests cardiac ejection fraction ≥50%;
   2. Serum creatinine ≤2.0× ULN, or creatinine clearance ≥60ml/min (CockcroftGault formula);
   3. ALT and AST≤3.0×ULN (≤5.0×ULN for patients with liver invasion);
   4. Total bilirubin ≤1.5 ×ULN (total bilirubin ≤3.0 ×ULN in Gilbert syndrome);
   5. Blood oxygen saturation ≥92% in non-oxygen state;
   6. Blood routine: neutrophils ≥1.0×109/L, platelets ≥75×109/L, hemoglobin ≥80g/L (with bone marrow invasion, neutrophils ≥0.5×109/L, platelets ≥50×109/L).
10. No serious mental disorders;
11. The venous access required for collection can be established, and mononuclear cell collection can be performed according to the judgment of the researcher, and there are no contraindications for other cell collection;
12. Women of childbearing age who have had a negative pregnancy test and all subjects agree to use a reliable and effective contraceptive method for contraception (excluding safe period contraception) for 1 year from signing the informed consent to receiving the infusion of MC-1-50 cells. Including but not limited to: abstinence, can inhibit ovulation implantable progesterone contraceptive; Intrauterine device (IUD); Intrauterine hormone release system; Spousal vasectomy; Combined hormonal contraceptives (oral, vaginal, and transdermal) that inhibit ovulation; Progesterone contraceptives (oral or injectable) that inhibit ovulation; Male subjects who have sex with a fertile female must consent to the use of a barrier method of contraception (e.g., condom plus spermicidal foam/gel/film/emulsion/suppository). At the same time, the subject should promise not to donate eggs (egg cells, oocytes) or sperm for assisted reproduction within 1 year after the cell infusion.

Exclusion Criteria:

1. Secondary CNS lymphoma was allowed to be included, except those with active CNS invasion or symptoms of CNS involvement or primary CNS lymphoma at the time of screening;
2. Patients who have received CAR-T therapy or other gene-modified cell therapy before screening;
3. Received allogeneic hematopoietic stem cell transplantation (allo-HSCT) before screening;
4. Received the following anti-tumor therapy before cell infusion: received chemotherapy, targeted therapy and other drug treatment (preconditioning) within 14 days or at least 5 half-lives (whichever is longer)

   Except for therapy and sheath chemotherapy for CNS lymphoma, which should be stopped 1 week before cell infusion); Received radiation within 14 days;
5. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA detection greater than the normal range; Hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA detection greater than the normal range; Positive for human immunodeficiency virus (HIV) antibodies; Syphilis positive; Cytomegalovirus (CMV) DNA test positive;
6. Have any of the following heart conditions:

   1. New York Heart Association (NYHA) Stage III or IV congestive heart failure;
   2. Had myocardial infarction or coronary artery bypass grafting (CABG) within 6 months prior to enrollment;
   3. A history of clinically significant ventricular arrhythmia, or unexplained syncope (other than those caused by vasovagal or dehydration);
   4. History of severe non-ischemic cardiomyopathy;
7. Active or uncontrollable infection requiring systemic treatment exists within 1 week prior to screening;
8. Grade 2 to 4 acute graft-versus-host disease (GVHD) or moderate to severe chronic GVHD were present within 4 weeks prior to screening;
9. Cerebrovascular accident or seizure occurred within 6 months before screening;
10. Occurrence of deep vein or deep artery embolization events within 6 months before screening;
11. Poor control of hypertension at screening, defined as systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg (blood pressure values are measured based on the average of 3 readings taken at least 2 minutes apart

    Patients with blood pressure ≥160/100mmHg at the initial screening can receive antihypertensive treatment, and if the blood pressure is well controlled after treatment and the blood pressure < 160/100mmHg can be screened);
12. Known to have active or uncontrolled autoimmune diseases, such as Crohns disease, rheumatoid arthritis, systemic lupus erythematosus, systemic vasculitis, etc., except skin diseases that do not require systemic treatment (e.g. Psoriasis);
13. Screening for interstitial lung disease requiring treatment;
14. Malignant tumors other than B-cell non-Hodgkin's lymphoma (except tumors with no active lesion and after treatment > 2 years, and adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, ductal carcinoma in situ after radical surgery);
15. Received live attenuated vaccine within 4 weeks prior to screening;
16. Participated in other interventional clinical studies within 4 weeks or 5 half-lives prior to screening;
17. Women who are pregnant or breastfeeding, as well as male or female subjects who plan to have a family within 1 year after receiving MC-1-50 cell transfusion;
18. Circumstances deemed unsuitable for participation in the study by other researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-12-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 1 month
  The incidence of adverse events after CAR-T cell infusion was assessed by the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 5.0)
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 1month
  Dose-limiting toxicity after CD19 CAR-T cell infusion

SECONDARY OUTCOMES:
Assessing objective response rate(ORR) of CAR-T cell preparations in CD19-positive relapsed/refractory B-cell non-Hodgkin lymphoma[Effectiveness] | 3 months
  Objective response rate after infusion 1 month and 3 month: The proportion of subjects who achieved CR, PR after CAR-T infusion accounted for all treated subjects (Assessed by investigators according to the Lugano 2014 criteria)#the minimum value is 0%#maximum value is 100%, and higher scores mean a better outcome.
Assessing best overall response rate(BOR) of CAR-T cell preparations in CD19-positive relapsed/refractory B-cell non-Hodgkin lymphoma[Effectiveness] | 3 months
  Best overall response rate rate after infusion 1 month and 3 month: proportion of patients who achieve optimal response (CR or PR) with MC-1-50 cell therapy (Assessed by investigators according to the Lugano 2014 criteria)#the minimum value is 0%#maximum value is 100%, and higher scores mean a better outcome.
Assessing best complete response rate(CRR) of CAR-T cell preparations in CD19-positive relapsed/refractory B-cell non-Hodgkin lymphoma[Effectiveness] | 3 months
  Complete response rate rate after infusion 1 month and 3 month: proportion of patients who achieve CR with MC-1-50 cell therapy (Assessed by investigators according to the Lugano 2014 criteria)#the minimum value is 0%#maximum value is 100%, and higher scores mean a better outcome.
Assessing best partial response rate(PRR) of CAR-T cell preparations in CD19-positive relapsed/refractory B-cell non-Hodgkin lymphoma[Effectiveness] | 3 months
  Partial response rate rate after infusion 1 month and 3 month: proportion of patients who achieve PR with MC-1-50 cell therapy (Assessed by investigators according to the Lugano 2014 criteria)#the minimum value is 0%#maximum value is 100%, and higher scores mean a better outcome.
AUCS of MC-1-50 cell preparation [Cell dynamics] | 3 months
  AUCS is defined as the area under the curve in 90 days
CMAX of MC-1-50 cell preparation [Cell dynamics] | 3 months
  CMAX is defined as the highest concentration of CEA CAR-T cells expanded in peripheral blood
TMAX of MC-1-50 cell preparation[Cell dynamics] | 3 months
  TMAX is defined as the time to reach the highest concentration
Pharmacodynamics of MC-1-50 cell preparation[Cell dynamics] | 3 months
  The clearance degree of CD19-positive B cells in peripheral blood was detected by flow cytometry at the visit points specified in the research protocol
To evaluate the immunogenicity positive rate of MC-1-50 cell preparation after infusion | 3 months
  The anti-CAR antibody was detected by ELISAt the visit points specified in the research protocol

OTHER OUTCOMES:
Objective response rate (ORR) of MC-1-50 cell treatment in patients with CD19-positive relapsed/refractory B-cell non-Hodgkin lymphoma[Effectiveness] | 2 years
  Objective response rate : The proportion of subjects who achieved CR, PR after CAR-T infusion accounted for all treated subjects (Assessed by investigators according to the Lugano 2014 criteria)#the minimum value is 0%#maximum value is 100%, and higher scores mean a better outcome.
Duration of Response (DOR) of MC-1-50 cell treatment in patients with CD19-positive relapsed/refractory B-cell non-Hodgkin lymphoma[Effectiveness] | 2 years
  DOR will be assessed from the first assessment of CR/PR to the first assessment of recurrence or progression of the disease or death from any cause
Progress-free survival(PFS) of MC-1-50 cell treatment in patients with CD19-positive relapsed/refractory B-cell non-Hodgkin lymphoma[Effectiveness] | 2 years
  PFS will be assessed from the first MC-1-50 cell infusion to death from any cause or the first assessment of progression
Overall survival(OS)of MC-1-50 cell treatment in patients with CD19-positive relapsed/refractory B-cell non-Hodgkin lymphoma[Effectiveness] | 2 years
  OS will be assessed from the first MC-1-50 cell infusion to death from any cause
Event-Free survival(EFS) of MC-1-50 cell treatment in patients with CD19-positive relapsed/refractory B-cell non-Hodgkin lymphoma[Effectiveness] | 2 years
  EFS will be assessed from the first MC-1-50 cell infusion to death from any cause or Disease progression or Treatment failure

CONTACTS AND LOCATIONS:
Overall Officials: Yuqin Song, M.D, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China